CLINICAL TRIAL: NCT05396105
Title: A Phase II/III, Extension Study of Orally Administered PHA-022121 for Acute Treatment of Angioedema Attacks in Patients With Hereditary Angioedema
Brief Title: Extension Study of Oral PHA-022121 for Acute Treatment of Angioedema Attacks in Patients With Hereditary Angioedema
Acronym: RAPIDe-2
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pharvaris Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHA022121-C303; 2023-505766-28-00 (EU CTIS Number)
Record Dates: First submitted 2022-04-28; First posted 2022-05-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Angioedema; Hereditary Angioedema Type I; Hereditary Angioedema Type II; Hereditary Angioedema Types I and II; Hereditary Angioedema Attack; Hereditary Angioedema With C1 Esterase Inhibitor Deficiency; Hereditary Angioedema - Type 1; Hereditary Angioedema - Type 2; C1 Esterase Inhibitor [C1-INH] Deficiency; C1 Esterase Inhibitor Deficiency; C1 Esterase Inhibitor, Deficiency of; C1 Inhibitor Deficiency; Hereditary Angioedema Type III; Hereditary Angioedema (HAE); Hereditary Angioedema Type I and II
Keywords: HAE; HAE Type I; HAE Type II; Oral Treatment; Bradykinin B2 Receptor Antagonists; On-Demand; PHA121; PHVS416; PHA-022121; Deucrictibant; HAE Type III
MeSH Terms: conditions — Angioedemas, Hereditary; Hereditary Angioedema Types I and II; Hereditary Angioedema Type III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Part B: Selected dose (Experimental): Single dose of deucrictibant
  Interventions: Drug: deucrictibant selected dose

INTERVENTIONS:
Drug: deucrictibant selected dose — deucrictibant soft capsule for oral use
  Other Names: PHVS416; PHA121; PHA-022121

SUMMARY:
This study evaluates the safety and efficacy of long-term on-demand treatment with orally administered deucrictibant for acute hereditary angioedema (HAE) attacks, including laryngeal attacks. The study will enroll patients from Study PHA022121-C201 (NCT04618211) and Study PHA022121-C306 (NCT06343779) who elect to participate in this extension study and meet the eligibility requirements.

DETAILED DESCRIPTION:
Part A of the study will enroll adult participants from Study PHA022121-C201. The double-blind treatment assignment from Study PHA022121-C201 will be maintained.

Part B will include participants rolling over from Part A and additionally enroll participants from Study PHA022121-C201 who did not participate in Part A, and participants from Study PHA022121-C306 who elect to participate in this extension study and meet the eligibility requirements.

ELIGIBILITY:
Key Inclusion Criteria:

1. Provision of written informed consent. If the participant is a minor (i.e., <18 years of age or as determined by local law), consent will be obtained from the participant's parent/legally designated representative/guardian and written assent will be obtained from the participant, per country regulations.
2. For participants from Study C201, received at least one dose of study drug (including the non-attack visit) in Study C201. For participants from Study C306, participant was randomized (and for adolescent participants 12 to <18 years received a dose of study drug in a non-attack state at Visit 1) and completed Study C306, with 2 attacks treated, or after closure of that study by the Sponsor.

   Enrollment of adolescents (≥12 to <18 years or age of adulthood as defined locally) from these studies is with consideration of local age requirements.
3. Female participants of childbearing potential (or who become of childbearing potential during the study) must agree to the protocol-specified pregnancy testing and to be abstinent from heterosexual intercourse or to use an acceptable contraception method as defined in the protocol and as available locally from enrollment until 30 days after the last study drug administration.
4. In the opinion of the Investigator, the participant (and parent/caregiver for adolescent participants) is willing and able to comply with the protocol.

Key Exclusion Criteria:

1. Any female who is pregnant, plans to become pregnant, or is breast-feeding.
2. Any other systemic disease (e.g., cardiovascular, gastrointestinal, renal, respiratory, neurological) or significant disease or disorder that, in the opinion of the Investigator, would interfere with the participant's safety or ability to participate in the study.
3. Use of lanadelumab for long-term HAE prophylactic therapy within 12 weeks prior to enrollment in Part A.
4. For Part A: Use of C1-esterase inhibitor, oral kallikrein inhibitors, attenuated androgens, anti-fibrinolytics, or monoclonal HAE therapy within a defined period prior to enrolment.

   For Part B: If a participant is receiving long-term prophylactic therapy with one of the following medications indicated for HAE: plasma-derived C1-INH, danazol at less than or equal to 200 mg/day, anti-fibrinolytics, berotralstat, or lanadelumab, they must be on a stable dose and regimen for at least 3 months before screening and intends to remain on the same dose for the duration of the study.
5. History of alcohol or drug abuse within defined period, or current evidence of substance dependence or abuse
6. Participation in any other investigational drug study within defined period
7. Discontinued from parent study after enrollment for any study drug-related safety reason or non-compliance including significant protocol deviation.
8. Use of concomitant medications that are strong CYP3A4 inhibitors (e.g., clarithromycin, erythromycin, itraconazole, ketoconazole, ritonavir) or strong CYP3A4 inducers (e.g., carbamazepine and phenytoin).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events (TEAEs), treatment-related TEAEs, treatment-emergent serious adverse events (TESAEs), treatment-related TESAEs, and TEAEs leading to deucrictibant discontinuation | From enrollment through study completion, up to 54 months (dependent on time of enrollment).
Heart Rate | From enrollment through study completion, up to 54 months (dependent on time of enrollment).
  Descriptive in nature, no formal statistical hypothesis testing will be performed.
Blood pressure | From enrollment through study completion, up to 54 months (dependent on time of enrollment).
  Systolic and diastolic blood pressure will be measured. Descriptive in nature, no formal statistical hypothesis testing will be performed.
Body temperature | From enrollment through study completion, up to 54 months (dependent on time of enrollment).
  Descriptive in nature, no formal statistical hypothesis testing will be performed.
Clinical laboratory tests | From enrollment through study completion, up to 54 months (dependent on time of enrollment).
  hematology, blood chemistry, urinalysis
Electrocardiograms | From enrollment through study completion, up to 54 months (dependent on time of enrollment).
Physical Examination | From enrollment through study completion, up to 54 months (dependent on time of enrollment).

SECONDARY OUTCOMES:
Time to onset of symptom relief, defined as Patient Global Impression of Change (PGI-C) rating of at least "a little better" for 2 consecutive timepoints within 12 hours post-treatment | Assessed from 1 hour to 12 hours post-treatment
  PGI-C evaluates the change in the attack symptoms over time with a 7-point response scale.
Time to substantial symptom relief, defined as achieving PGI-C rating of at least "better" for 2 consecutive timepoints within 12 hours post-treatment | Assessed from 1 hour to 12 hours post-treatment
  PGI-C evaluates the change in the attack symptoms over time with a 7-point response scale.
Time to substantial symptom relief by Patient Global Impression of Severity (PGI-S), defined as achieving ≥1 point reduction in PGI-S from pre-treatment for 2 consecutive timepoints within 12 hours post-treatment | Assessed from pre-treatment to 12 hours post-treatment
  PGI-S evaluates the severity of attack symptoms with a 5-point response scale.
Time to onset of symptom relief by VAS-3/VAS-5 (Part A) or AMRA (Part B), defined as a reduction of ≥30% from pretreatment in VAS/AMRA composite score, sustained for 2 consecutive timepoints) | Assessed from pre-treatment to 48 hours post-treatment
  VAS scores range between 0 and 100. A larger reduction means a better outcome.
Time to symptom relief by VAS (Part A) or AMRA (Part B), based on achieving ≥50% reduction from pretreatment in VAS/AMRA composite score sustained for 2 consecutive timepoints. | Assessed from pre-treatment to 48 hours post-treatment
  VAS/AMRA scores range between 0 and 100. A larger reduction means a better outcome.
Proportion of deucrictibant-treated attacks requiring rescue medication within 24 hours post-treatment | Assessed from pre-treatment to 24 hours post-treatment
Proportion of deucrictibant-treated attacks with almost complete or complete symptom relief by VAS-3/ VAS-5/ AMRA through 24 hours post-treatment | Assessed from pre-treatment to 24 hours post-treatment
  Almost complete or complete symptom relief is defined as all individual item scores in VAS/AMRA having a value ≤10 sustained for 2 consecutive timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Pharvaris Netherlands B.V.
Locations (57):
- United States (13):
  - Study site, Birmingham, Alabama
  - Study site, Scottsdale, Arizona
  - Study site, Little Rock, Arkansas
  - Study site, San Diego, California
  - Study site, Santa Monica, California
  - Study site, Walnut Creek, California
  - Study site, Colorado Springs, Colorado
  - Study site, Chevy Chase, Maryland
  - Study site, Boston, Massachusetts
  - Study site, Detroit, Michigan
  - Study site, St Louis, Missouri
  - Study site, Hershey, Pennsylvania
  - Study site, Dallas, Texas
- Argentina (2):
  - Study site, Buenos Aires
  - Study site, Salta
- Study site, Campbelltown, New South Wales, Australia
- Austria (2):
  - Study site, Graz
  - Study site, Vienna
- Brazil (4):
  - Study site, Salvador, Estado de Bahia
  - Study site, Ribeirão Preto
  - Study site, Santo André
  - Study site, São Paulo
- Study site, Sofia, Bulgaria
- Canada (2):
  - Study site, Edmonton, Alberta
  - Study site, Montreal, Quebec
- Study site, Brno, Czechia
- France (2):
  - Study site, Grenoble
  - Study site, Paris
- Germany (3):
  - Study site, Berlin
  - Study site, Frankfurt am Main
  - Study site, Lübeck
- Study site, Hong Kong, Hong Kong
- Study site, Budapest, Hungary
- Study site, Ashkelon, Israel
- Italy (6):
  - Study site, Catania
  - Study site, Milan
  - Study site, Napoli
  - Study site, Padua
  - Study site, Palermo
  - Study site, Roma
- Japan (4):
  - Study site, Hiroshima
  - Study site, Kanagawa
  - Study site, Osaka
  - Study site, Tokyo
- Study site, Amsterdam, Netherlands
- Study site, Krakow, Poland
- Study site, San Juan, Puerto Rico
- Study site, Riyadh, Saudi Arabia
- Study site, Cape Town, South Africa
- South Korea (2):
  - Study site, Daegu
  - Study site, Seoul
- Spain (2):
  - Study site, Barcelona
  - Study site, Madrid
- Study site, Lund, Sweden
- Turkey (Türkiye) (2):
  - Study site, Ankara
  - Study site, Istanbul
- Study site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No